CLINICAL TRIAL: NCT05031494
Title: A Multi-center, Open-label Phase II Study to Evaluate the Safety and Efficacy of YH003 in Combination with Toripalimab (anti-PD-1 MAb) in Patients with Unresectable/metastatic Melanoma and Pancreatic Ductal Adenocarcinoma (PDAC)
Brief Title: A Study to Assess YH003 in Combination with Toripalimab(anti-PD-1 MAb) Injection in Patients with Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eucure (Beijing) Biopharma Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YH003004
Record Dates: First submitted 2021-08-26; First posted 2021-09-02 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Melanoma; Pancreatic Ductal Adenocarcinoma
MeSH Terms: conditions — Melanoma | interventions — toripalimab; 130-nm albumin-bound paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- YH003 with Toripalimab in subjects with unresectable /metastatic melanoma (Experimental): YH003 in combination with Toripalimab in subjects with unresectable /metastatic melanoma after having failed PD-1/L1 +/- CTLA-4 treatment;
  Interventions: Drug: YH003; Drug: Toripalimab
- YH003 with Toripalimab in subjects with PDAC (Experimental): YH003 in combination with Toripalimab in subjects with unresectable/ metastatic pancreatic ductal adenocarcinoma (PDAC) as 2nd line treatment;
  Interventions: Drug: YH003; Drug: Toripalimab
- YH003 with Toripalimab plus standard chemotherapy (Experimental): YH003 in combination with Toripalimab plus standard chemotherapy (Nab-paclitaxel + Gemcitabine) in subjects with unresectable/metastatic PDAC as 1st line treatment;
  Interventions: Drug: YH003; Drug: Toripalimab; Drug: Nab-paclitaxel; Drug: Gemcitabine

INTERVENTIONS:
Drug: YH003 — YH003 will be dosed at RP2D every 3 weeks. The first infusion of YH003 should be administered over 60 minutes.
Drug: Toripalimab — Toripalimab will be administered at a dose of 240 mg every 3 weeks.
Drug: Nab-paclitaxel — Nab-paclitaxel will be administered each 21-day cycle.
  Arms: YH003 with Toripalimab plus standard chemotherapy
Drug: Gemcitabine — Gemcitabine will be administrated each 21-day cycle.
  Arms: YH003 with Toripalimab plus standard chemotherapy

SUMMARY:
A phase II, multi-center, open-label study to evaluate the safety and efficacy of YH003 in combination with Toripalimab (anti-PD-1 mAb) in patients with unresectable/metastatic melanoma and pancreatic ductal adenocarcinoma (PDAC)

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for study entry patients must satisfy all of the following criteria:
* 1. Subjects must have the ability to understand and willingness to sign a written informed consent document.
* 2. Histologically or cytologically confirmed unresectable or metastatic melanoma and pancreatic ductal adenocarcinoma
* Cohort 2A: had confirmed progressive disease during treatment with an anti-PD-1/PD-L1 with or without CTLA-4 therapy.
* Cohort 2B: had confirmed progressive disease during treatment with first line standard of care chemotherapy per local guideline.
* Cohort 2C: must not have received any prior systematic treatment, including chemotherapy, biological therapy, or targeted therapy for unresectable locally advanced/ metastatic pancreatic duct adenocarcinoma.
* 3. Subject must have at least 1 unidimensional measurable disease by RECIST 1.1.
* 4. Subjects must be age between 18 years.
* 5. Subjects must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* 6. Life expectancy ≥3 months.
* 7. Subjects must have adequate organ function

Exclusion Criteria:

* Subjects who meet any of the following criteria cannot be enrolled:
* 1. Cohort 2A: History of life-threatening toxicity or treatment discontinuation due to related to prior anti-PD-1/PD-L1 with or without CTLA-4 treatment for subjects with unresectable/ metastatic melanoma
* 2.Subjects have another active invasive malignancy within 5 years, with the following exceptions and notes:
* 3. Previous exposure to TNFR such as anti-CD137, OX40, CD27 and CD357 antibodies.
* 4. Subjects must not have received any anticancer therapy or another investigational agent within the shorter of 4 weeks or 5 half-lives before the first dose of the study treatment.
* 5. Subjects with a history of ≥ Grade 3 immune-related adverse events resulted from previous immunotherapy or treatment discontinuation due to previous immunotherapy. .
* 6. History of clinically significant sensitivity or allergy to monoclonal antibodies and their excipients or known allergies to antibodies produced from Chinese hamster ovary cells, which in the opinion of the Investigator suggests an increased potential for an adverse hypersensitivity to YH003 or Toripalimab. (For cohort 2C: history of severe hypersensitivity reaction to Nap-paclitaxel and/or gemcitabine).
* 7. Primary central nervous system (CNS) malignancies or symptomatic CNS metastases.
* 8. History of (non-infectious) pneumonitis that required corticosteroids or current pneumonitis, or history of interstitial lung disease.
* 9. Active, hemodynamically significant pulmonary embolism within 12 weeks prior to the first dose of study drug.
* 10. Subjects must not have a known or suspected history of an autoimmune disorder
* 11. Clinically uncontrolled intercurrent illness,
* 12. Severe cardiovascular disease including symptomatic congestive heart failure (New York Heart Association class III or IV), unstable angina, uncontrolled hypertension, cardiac arrhythmia, a history of myocardial infarction within 6 months or a history of arterial thromboembolic event and pulmonary embolism within 3 months of the first dose of investigational agent.
* 13. QTc > 480 ms (Fridericia equation) at baseline; no concomitant medications that would prolong the QT interval; no family history of long QT syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-12-08 (Actual); Primary Completion 2023-08-16 (Actual); Study Completion 2023-08-16 (Actual)

PRIMARY OUTCOMES:
Confirmed Objective Response Rate (ORR) | up to 1 year after the last dosing
  Overall Response Rate (ORR) by investigator's assessment according to the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1

SECONDARY OUTCOMES:
Adverse events (AE) | up to 1 year after the last dosing
  The safety profile of YH003 in combination with Toripalimab will be assessed by monitoring the adverse events (AE) per NCI CTCAE v5.0
Duration of response (DOR) | up to 1 year after the last dosing
  To assess the antitumor activity of YH003 in combination with Toripalimab
Time to response (TTR) | up to 1 year after the last dosing
  To assess the antitumor activity of YH003 in combination with Toripalimab
Progression free survival (PFS) | up to 1 year after the last dosing
  To assess the antitumor activity of YH003 in combination with Toripalimab
Disease control rate (DCR) | up to 1 year after the last dosing
  To assess the antitumor activity of YH003 in combination with Toripalimab
Duration of disease control (DDC) | up to 1 year after the last dosing
  To assess the antitumor activity of YH003 in combination with Toripalimab
Overall survival (OS) | up to 1 year after the last dosing
  To assess the antitumor activity of YH003 in combination with Toripalimab
Incidence of neutralizing antibodies (NAbs) | up to 1 year after the last dosing
  To assess the immunogenicity of YH003 in combination with Toripalimab

CONTACTS AND LOCATIONS:
Locations (2):
- Ichan School of Medicine at Mount Sinai, New York, New York, United States
- Epworth Medical Centre, Richmond, Victoria, Australia